CLINICAL TRIAL: NCT00664131
Title: Neurologic Morbidity and Disability in Acute Lymphoblastic Leukemia Survivors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ALLNOQ
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL survivors; ALL neurologic symptoms; ALL neurologic disability; ALL late effects
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Neurological Examination/Questionnaires

INTERVENTIONS:
Other: Neurological Examination/Questionnaires — See Detailed Description section for description of treatment plan.

SUMMARY:
Treatment of acute lymphoblastic leukemia achieves high cure rate, but is potentially neurotoxic.

Long-term neurologic morbidity in survivors and its effect on function are inadequately studied.

Neurologic outcomes will be assessed through an investigator administered questionnaire followed by comprehensive neurologic examination by the study neurologist.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is the most prevalent childhood malignant disease. Survival has improved from 5-10% in the early 1960s to over 80% at present. Historically, the central nervous system (CNS) was the most common site of leukemia relapse. However, major improvement in cure rates was achieved with the addition of CNS directed therapy using initially craniospinal irradiation, and more recently, a combination of high-dose systemic methotrexate and intrathecal chemotherapy.

ALL mostly afflicts children in the first 12-years of life, an age when progressive myelination is taking place and the central nervous system is more vulnerable to chemical and radiologic injury. Many ALL studies have reported neurologic adverse events related to the treatment.

Little is known about the long-term outcome of neurologic toxicity developing during treatment of leukemia, or development of new late onset neurologic complications. No data is available about outcomes of non-behavioral/cognitive neurologic complications, such as seizures, incoordination, headache, loss of motor or sensory function, impaired energy and muscle weakness. In addition, there is no data available on impact of neurologic disability on quality of life of ALL survivors.

It is important to understand and recognize neurologic disability, its causes and impact on function and quality of life so that adequate and timely remedies can be offered through education and appropriate interventions can be undertaken to help prevent long-term morbidity.

This is a prospective observational study of ALL St. Jude Children's Research Hospital survivors to determine the prevalence of different headache syndromes, as defined by International Society of Headache criteria (IHS) and the prevalence and severity of seizures and their relationship to leukemia treatment. We will establish incidence, type, severity, and disability of sensory-motor neuropathy when present or any long term progression of initial peripheral nerve injury in ALL survivors. This study will also help define whether there is a higher incidence of low back pain and if there is any relation to a specific treatment.

Subjects will have a one-time evaluation with an investigator administered questionnaire and a neurologic examination.

ELIGIBILITY:
Inclusion Criteria:

* Childhood ALL survivors treated on institutional protocols at
* Patient will be at least 5-years from ALL diagnosis.
* Patient will be at least one year from completion of cancer therapy.
* Absence of recurrent or secondary cancer for at least one year day of enrollment.
* Between 6-28 years of age at the time of evaluation.
* Patient's or at least one parent's English is proficient enough Questionnaire.
* Parent and the child agree to participate. Consent only from will suffice if > 18 years of age at the time of assessment.

Exclusion Criteria:

* Recurrent tumor or development of secondary cancer
* Child or parent refuses to participate
* Co-morbid pre-existing disabling neurologic disease, which in the judgment of the principal investigator may compromise clinical observations.

Ages: 6 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Survivors of ALL who are currently 6-28 years of age, 5 years from ALL diagnosis, and 1 year off therapy who were treated on institutional protocols at St. Jude Children's Research Hospital. Survivors will be recruited in the Leukemia and ACT clinics at St. Jude Children's Research Hospital. We anticipate that 494 survivors are available. We plan to enroll every survivor who is eligible and visits Leukemia or/ and ACT clinic at St. Jude Children's Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2005-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To estimate prevalence of neurologic symptoms as reported by the patient or parent in childhood acute lymphoblastic leukemia survivors. | At lease 5 years from diagnosis and at least one year after completion of therapy.
To estimate prevalence of neurologic signs as determined by detailed neurologic examination of childhood acute lymphoblastic leukemia survivors. | At lease 5 years from diagnosis and at least one year after completion of therapy.

SECONDARY OUTCOMES:
To estimate prevalence of neurologic disability as determined by neurologic symptoms, signs and administered questionnaire instruments. | At lease 5 years from diagnosis and at least one year after completion of therapy.
To explore risk factors for development of neurologic disability. | At lease 5 years from diagnosis and at least one year after completion of therapy.
To assess effect of neurologic disability on quality of life. | At lease 5 years from diagnosis and at least one year after completion of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Ness, PT, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org